CLINICAL TRIAL: NCT02343029
Title: Physical Activity and Cerebral Metabolism in the Elderly: a Randomised Controlled Trial
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Johannes Pantel (Other)
Responsible Party: Sponsor-Investigator, Professor Johannes Pantel, Head of Department, Institute of General Practice, Goethe University
Organization: Goethe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMART
Record Dates: First submitted 2015-01-12; First posted 2015-01-21 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Dementia; Cognitive Impairment
Keywords: Aerobic Exercise Training; prevention; magnetic resonance spectroscopic imaging; psychometric tests; cognition; dementia; cognitive impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in the Intervention group exercise three times a week for 30 minutes on a bicycle ergometer (optibike med, ergoline GmbH, Bitz, Germany) in the integrated gym hall of one of the participating residencies. Training is individualised as respective performance is adapted to the power at the first ventilator threshold (assessed during cardiopulmonary exercise test).
  Interventions: Other: Individualised aerobic exercise training
- Waiting Control (Active Comparator): Participants of Waiting Control continue their regular physical activity behaviour for 12 weeks. They will start the same exercise intervention after a reassessment at week 12 for the next upcoming 12 weeks. (13-24)
  Interventions: Other: Individualised aerobic exercise training; Other: Waiting Control

INTERVENTIONS:
Other: Individualised aerobic exercise training — During the first 4 weeks of intervention two of the three weekly training sessions are offered as group training supervised by the respective qualified exercise physiologist of the Department of Sports Medicine. After 4 weeks, participants' physical performance is reassessed at the Department of Sports Medicine. If necessary, workload is readjusted to achieve the initially defined exercise intensity.
Other: Waiting Control — After waiting for 12 weeks with normal daily activity, patients are allocated to a individualised aerobic exercise training, too.
  Arms: Waiting Control

SUMMARY:
Physical activity exerts a variety of long-term health benefits in older adults.This randomised controlled trial investigates the effect of a 12-week physical exercise program on the change in cerebral metabolism as assessed with Magnetic Resonance Spectroscopic Imaging. Follow-up lasts for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. be above 65 years of age,
2. voluntariness
3. capacity to consent,
4. having passed medical entry exam by the Department of Sports Medicine,

4) regular mental capacity, 5) written informed consent

Exclusion Criteria:

1. untreated clotting disorders,
2. musculoskeletal diseases significantly reducing mobility,
3. severe bacterial or viral infections,
4. severe respiratory diseases (Gold IV),
5. acute pulmonary embolism,
6. instable angina pectoris or severe heart failure (NYHA III or IV),
7. severe vascular disease of the extremities or the brain,
8. severe pulmonary-cardiac dysfunction,
9. acute myocardial infarction or early phase of rehabilitation,
10. critical aortal stenosis,
11. severe hypertrophic and obstructive cardiomyopathy,
12. untreated malignant arrhythmias,
13. untreated severe hypertonia,
14. severe pulmonary hypertonia,
15. symptomatic cardiac malformations,
16. cardiac-block grade II or III,
17. left bundle branch block,
18. complex ventricular arrhythmias,
19. Cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in cerebral metabolism (assessed by MRSI) | 6 month
  assessed by MRSI, Primary hypothesis is that aerobic exercise leads to an increase of cerebral N-acetyl-aspartate (NAA; mediated by plasma neurotrophins).
  Secondary hypothesis stipulates an increase of markers of neuronal energy reserve: i.e. the ratio of phosphocreatinin to creatinine and of adenosine-tri-phosphate (ATP) to ~di-phosphate (ADP).
  Third hypothesis is an increase in the volume of cortical grey matter

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (Aerobic exercise capacity is determined by a physician-supervised CPET) | 0, 3 and 6 month
  Aerobic exercise capacity is determined by a physician-supervised CPET
Psychometric testing 1 (verbal declarative memory [Verbal Learning and Memory test; adapted German version of the Rey Auditory Verbal Learning test] | 0, 3 and 6 month
  verbal declarative memory [Verbal Learning and Memory test; adapted German version of the Rey Auditory Verbal Learning test]
Psychometric testing 2 (frontal executive control [Colour-Word-Interference test; adapted German version of the Stroop test; Trail-Making-Test Part B] | 0, 3 and 6 month
  frontal executive control [Colour-Word-Interference test; adapted German version of the Stroop test; Trail-Making-Test Part B]
Psychometric testing 3 (working memory [Digit Span Test forward and backward] | 0, 3 and 6 month
  working memory [Digit Span Test forward and backward]
Psychometric testing 4 9semantic and phonematic fluency, nonverbal declarative memory and visual-constructive abilities by means of the CERAD-Plus (Consortium to Establish a Registry for Alzheimer's Disease) Neuropsychological Battery) | 0, 3 and 6 month
  semantic and phonematic fluency, nonverbal declarative memory and visual-constructive abilities by means of the CERAD-Plus (Consortium to Establish a Registry for Alzheimer's Disease) Neuropsychological Battery
Psychometric testing 5 (speed of cognitive processing is assessed by means of the Trail-Making-Test Part A) | 0, 3 and 6 month
  speed of cognitive processing is assessed by means of the Trail-Making-Test Part A
Psychometric testing 6 (depressive disorders: Geriatric Depression Scale) | 0, 3 and 6 month
  depressive disorders: Geriatric Depression Scale
Psychometric testing 7 (Age-associated subjective memory impairment is assessed using a memory complaint questionnaire [MAC-Q] | 0, 3 and 6 month
  Age-associated subjective memory impairment is assessed using a memory complaint questionnaire [MAC-Q]
Psychometric testing 8 (cristalline intelligence is assessed by means of a verbal intelligence test [Multiple-Choice Word Test: MWT-B] | 0, 3 and 6 month
  cristalline intelligence is assessed by means of a verbal intelligence test [Multiple-Choice Word Test: MWT-B]
Psychometric testing 9 (dementia and mild cognitive impairment using the Mini Mental State Examination and the Instrumental Activities of Daily Living Questionnaire) | 0, 3 and 6 month
  dementia and mild cognitive impairment using the Mini Mental State Examination and the Instrumental Activities of Daily Living Questionnaire
Balance and strength (postural sway (balance) and gait data acquisition via the capacitive force-measuring platform (30 Hz) WinFDM v0.0.41® (Zebris© GmbH, Isny, Germany) | 0, 3 and 6 month
  postural sway (balance) and gait data acquisition via the capacitive force-measuring platform (30 Hz) WinFDM v0.0.41® (Zebris© GmbH, Isny, Germany)
Pain Assessment (German Pain Questionnaire) | 0, 3 and 6 month
  German Pain Questionnaire
History of diet (Food frequency questionnaire DEGS1) | 0, 3 and 6 month
  Food frequency questionnaire DEGS1
History and fear of falling (German version of the Falls-Efficacy-Scale International Version) | 0, 3 and 6 month
  German version of the Falls-Efficacy-Scale International Version
Physical activity (International Physical Activity Questionnaire, Lifetime Total Physical Activity Questionnaire and Accelerometry) | 0, 3 and 6 month
  International Physical Activity Questionnaire, Lifetime Total Physical Activity Questionnaire and Accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Pantel, Prof., Principal Investigator — Institute of General Practice, Goethe University, Frankfurt/Main, Germany; Winfried E Banzer, Prof., Principal Investigator — Department of Sports Medicine, Institute of Sports Sciences, Goethe University, Frankfurt/Main, Germany
Locations (2):
- Germany (2):
  - Department of Sports Medicine, Institute of Sports Sciences, Goethe University, Frankfurt am Main
  - Institute of General Practice, Goethe University,, Frankfurt am Main

REFERENCES:
- [Background] Fleckenstein J, Matura S, Engeroff T, Fuzeki E, Tesky VA, Pilatus U, Hattingen E, Deichmann R, Vogt L, Banzer W, Pantel J. SMART: physical activity and cerebral metabolism in older people: study protocol for a randomised controlled trial. Trials. 2015 Apr 11;16:155. doi: 10.1186/s13063-015-0662-9. PMID 25872789